CLINICAL TRIAL: NCT05864417
Title: A Single-Center, Open-Label, Safety in Use Clinical Study to Assess Topical Tolerability and Efficacy in Improving Wrinkles, Fine Lines, and Melasma After 84 ± 2 Days of Use of Two Facial Sunscreens in Adult Participants
Brief Title: A Study to Assess Effect of Two Facial Sunscreens in Improving Wrinkles, Fine Lines and Melasma in Adult Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA005235; CCSSKA005235 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunscreen (Experimental): Participants will choose one facial sunscreen (SPF 70) out of the two (one with a light tone [Color 2.0] and another with a medium tone [Color 3.0]) based on the tone that best suits their skin color. At home, they will apply a generous amount of facial sunscreen to the face twice daily and will reapply when they feel the need up to 84 + (-) 2 days.
  Interventions: Other: Sunscreen Color tone 2.0; Other: Sunscreen Color tone 3.0

INTERVENTIONS:
Other: Sunscreen Color tone 2.0 — Participants will topically apply sunscreen color tone 2.0.
Other: Sunscreen Color tone 3.0 — Participants will topically apply sunscreen color tone 3.0.

SUMMARY:
The purpose of this study is to evaluate the topical safety (tolerability/acceptability) and efficacy of two facial sunscreen in improving wrinkles, fine lines and melasma after 84 +/- 2 days of use under normal conditions on the face by adult participants. For these investigational products, safety parameters, clinical efficacy, instrumental efficacy (assessment of color intensity and size of melasma spots and assessment of wrinkles and fine lines), facial imaging, and self-perceived efficacy through subjective questionnaire and quality of life questionnaires (MELASQol) will be evaluated, as well as an open emotional statement written by the participant at the end of use experience".

ELIGIBILITY:
Inclusion Criteria:

* Male and/or Female
* Participants of any ethnicity according to IBGE criteria
* From 35 years of age
* Fitzpatrick Skin Type II to IV
* Participant presenting mild to moderate melasma (grade 1 to 2 - according to the Site's scale), proven by a dermatologist
* Participant's presenting wrinkles/fine lines in any region of the face (periorbital, frontal and/or nasolabial) from grade 2 to 6 (according to the Site's scale), confirmed by the dermatologist
* Generally in good health based on medical history reported by the participant
* Able to read, write, speak, and understand Portuguese
* For Male Participants: agree to shave 24 hours before visits 1 to 4
* Individual has signed the following informed consent documents (ICD):ICD, Informed Consent Image Disclosure (ICID) e Informed Consent for Cession of Rights for Image Use (ICCRIU)
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products including sunscreen
* Presents with a skin condition that may confound the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer)
* Presents with primary/secondary lesions (example scars, ulcers, vesicles) or tattoos on test sites
* Participants with immune deficiency
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including - immunosuppressive or steroidal drugs within 2 months before Visit 1, 2; non-steroidal anti-inflammatory drugs within 5 days before Visit 1; antihistamines within 2 weeks before Visit 1
* Start or change of hormone replacement therapy or contraceptive drug method in the last 03 months
* Participants who are using or have used topical products such as Retin-A, Retin-A Micro, and Differin or any other topical retinoid on the face within 6 months prior to the study; or use of any oral retinoid within 1 year prior to the study
* Participants who are using or have currently used any facial products containing active ingredients against spots and/or wrinkles: alpha or beta hydroxy acids (including salicylic acid), polyhydroxy acids, topical products containing retinol or retinol derivatives, hydroquinones, arbutin, niacinamide, N-acetylglucosamine, Thiamidol, kojic acid, azelaic acid, licorice extract, whitening peptides, vitamin C or any other 'anti-aging' products or products capable of interfering with skin brightness/uniformity, or with spots, within 2 months prior to the start of the study
* Participants who have used cosmetic products on the same area (face) with anti-spot and anti-wrinkle action, within 14 days before the beginning of the study
* Participants who have undergone chemical and/or physical peeling, laser or similar aesthetic treatments within 6 months prior to the study
* Participants who have undergone invasive cosmetic or dermatological treatment in the test area within 2 months before the start of the study or during the study
* Intense sun exposure or tanning session up to 01 month before the initial evaluation or planned intense sun exposure or tanning session during the study
* Present signs of intense tanning, according to the evaluation of the study physician
* Is self-reported to be pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Present excessive hair in the evaluation region that may interfere in the instrumental measurements. In the case of men, even in the presence of excessive hair in the beard region, they will be instructed to shave one day before the visit
* Is simultaneously participating in any other clinical study;
* Is an employee/contractor or immediate family member of the principal investigator (PI), Study Site, or Sponsor

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 84 +/- 2 days
  Number of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/ frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.
Improvement in Assessment of Melasma Color Intensity Using Chroma Meter CR 400 at Day 28 | Baseline and Day 28
  Melasma color intensity will be measured using chroma meter. Measurements will be performed both in area with melasma chosen by dermatologist, as documented in CRF during the eligibility assessment, and in an adjacent region (without the presence of melasma). Statistical improvement will be measured as (reduction in value of "b" parameter and increase in value of "L" and ITA parameters) versus baseline (D1) and Day 28 by an Anova model followed by Fisher's least significant difference (LSD) multiple comparison test. The color space L *, a *, b * was developed as a method of expressing colors in terms of numbers. The color space corresponds to perceived color characterization. L * stands for brightness (100 corresponds to white and 0 corresponds to black and b * indicates blue-yellow coloration. By determining values L * and b * of a color, it is possible to calculate individual topology angle (ITA). The lighter the skin, the higher the ITA.
Improvement in Assessment of Melasma Color Intensity Using Chroma Meter CR 400 at Day 56 | Baseline and Day 56
  Melasma color intensity will be measured using chroma meter. Measurements will be performed both in area with melasma chosen by dermatologist, as documented in CRF during the eligibility assessment, and in an adjacent region (without the presence of melasma). Statistical improvement will be measured as (reduction in value of "b" parameter and increase in value of "L" and ITA parameters) versus baseline (D1) and Day 28 by an Anova model followed by Fisher's LSD multiple comparison test. The color space L *, a *, b * was developed as a method of expressing colors in terms of numbers. The color space corresponds to perceived color characterization. L * stands for brightness (100 corresponds to white and 0 corresponds to black and b * indicates blue-yellow coloration. By determining values L * and b * of a color, it is possible to calculate ITA (individual topology angle). The lighter the skin, the higher the ITA.
Improvement in Assessment of Melasma Color Intensity Using Chroma Meter CR 400 at Day 84 +/- 2 | Baseline and Day 84 +/- 2
  Melasma color intensity will be measured using chroma meter. Measurements will be performed both in area with melasma chosen by dermatologist, as documented in CRF during the eligibility assessment, and in an adjacent region (without the presence of melasma). Statistical improvement will be measured as (reduction in value of "b" parameter and increase in value of "L" and ITA parameters) versus baseline (D1) and Day 28 by an Anova model followed by Fisher's LSD multiple comparison test. The color space L *, a *, b * was developed as a method of expressing colors in terms of numbers. The color space corresponds to perceived color characterization. L * stands for brightness (100 corresponds to white and 0 corresponds to black and b * indicates blue-yellow coloration. By determining values L * and b * of a color, it is possible to calculate ITA (individual topology angle). The lighter the skin, the higher the ITA.
Number of Participants with Improvement From Baseline in Melasma, and Wrinkles and Fine lines Assessed Using the Visia-CR Facial Imaging Booth at Day 28 | Baseline and Day 28
  Facial images will be captured using the Visia CR Facial Imaging Booth. Three images per participant will be captured: right lateral, left lateral and frontal using the Standard 1, Standard 2, Cross Polarized and RBX (Brown) filters.The captured images will be further analyzed using specific image analysis software to evaluate the intensity and size of melasma, and wrinkles and fine lines.
Number of Participants with Improvement From Baseline in Melasma, and Wrinkles and Fine lines Assessed Using the Visia-CR Facial Imaging Booth at Day 56 | Baseline and Day 56
  Facial images will be captured using the Visia CR Facial Imaging Booth. Three images per participant will be captured: right lateral, left lateral and frontal using the Standard 1, Standard 2, Cross Polarized and RBX (Brown) filters.The captured images will be further analyzed using specific image analysis software to evaluate the intensity and size of melasma, and wrinkles and fine lines.
Number of Participants with Improvement From Baseline in Melasma, and Wrinkles and Fine lines Assessed Using the Visia-CR Facial Imaging Booth at Day 84 +/- 2 | Baseline and Day 84 +/- 2
  Facial images will be captured using the Visia CR Facial Imaging Booth. Three images per participant will be captured: right lateral, left lateral and frontal using the Standard 1, Standard 2, Cross Polarized and RBX (Brown) filters.The captured images will be further analyzed using specific image analysis software to evaluate the intensity and size of melasma, and wrinkles and fine lines.
Number of Participants With Improvement From Baseline in Quality of Life as Assessed by the Melasma Quality of Life Scale (MELASQOL) at Day 28 | Day 28
  The MELASQol assesses the effect melasma has on the quality of life of sufferers on a scale of 1-10, where 1=not bothered at all, 2=not bothered most of the time,3=not bothered sometimes,4= neutral,5=sometimes bothered,6=Mostly bothered and 7=bothered all the time to 7 (bothered all of the time) rating the 10 questions. A total score is generated which ranges from 10 to 70. The lower the score, the better the participant's quality of life.
Number of Participants With Improvement From Baseline in Quality of Life as Assessed by the Melasma Quality of Life Scale (MELASQOL) at Day 56 | Day 56
  The MELASQol assesses the effect melasma has on the quality of life of sufferers on a scale of 1-10, where 1=not bothered at all, 2=not bothered most of the time,3=not bothered sometimes,4= neutral,5=sometimes bothered,6=Mostly bothered and 7=bothered all the time to 7 (bothered all of the time) rating the 10 questions. A total score is generated which ranges from 10 to 70. The lower the score, the better the participant's quality of life.
Number of Participants With Improvement From Baseline in Quality of Life as Assessed by the Melasma Quality of Life Scale (MELASQOL) at Day 84 +/- 2 | Day 84 +/- 2
  The MELASQol assesses the effect melasma has on the quality of life of sufferers on a scale of 1-10, where 1=not bothered at all, 2=not bothered most of the time,3=not bothered sometimes,4= neutral,5=sometimes bothered,6=Mostly bothered and 7=bothered all the time to 7 (bothered all of the time) rating the 10 questions. A total score is generated which ranges from 10 to 70. The lower the score, the better the participant's quality of life.
Participant's Self-perceived Questionnaire to Assess their Perception of the Color/Tone of Sunscreen | Baseline (Day 1)
  Participants will apply the investigational products on their faces, one product on each half-face to see how the color of each product will look in relation to their skin tone, and then choose the product that best suits their skin color.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 28 | Day 28
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 28 will be reported. Participants will answer 3 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 84 +/- 2 | Day 84 +/- 2
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 84 +/- 2 will be reported. Participants will answer 14 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.
Testimonial Regarding the Experience with Sunscreen | End of the Study (84 +/- 2 days)
  A testimonial regarding the experience with sunscreen will be provided by the participants through an open question at the end of the study. The purpose is to know their opinion and experience using this product during the study.
Topical Tolerability as Assessed by the Dermatologist | Up to 84 +/- 2 days
  Topical tolerability will be assessed using skin reaction intensity evaluation scale. Skin Reaction Intensity Evaluation Scale is a composite evaluation of any irritation/reaction subscoring for erythema, peeling, vesiculation, and edema. The scale ranges from 0=absent to 4=intense.
Number of Participants with Improvement From Baseline in Melasma by mMASI Scale as Assessed by the Dermatologist | Up to 84 +/- 2 days
  The modified mMASI scale (Area and Severity Index) will be used. The evaluation is performed under standard lighting (day light). The modified mMASI scale score is calculated by subjectively assessing two factors: area of involvement (A) and darkening (D), with the forehead (f), right malar region (rm), left malar region (lm), and chin (c), corresponding to 30%, 30%, 30%, and 10% of the total face, respectively. The grading range is from 0 to 24, and the area of involvement (A) and darkening (D) are graded as described below:Area of Involvement (A): 0= absent, 1 = <10%, 2 = 10%-29%, 3 = 30%-49%, 4 = 50%-69%, 5 = 70%-89%, 6 = 90%-100% and Darkening (D):0= absent, 1 = very light, 2 = light, 3= significantly, 4 = severe.
Clinical Efficacy Evaluations as Assessed by the Dermatologist on Day 28 | Day 28
  It is a clinical evaluation of the participant's face performed by a dermatologist according to a predefined scale. The attributes evaluated will be: wrinkles, and fine lines. A 10-point ordinal scale (0 to 9) developed by study site will be used where 0 = Absent and 9 = Numerous.Therefore, because it is an ordinal scale, the points in between do not have an established definition.
  Dermatologists have been trained to evaluate and classify grades 1, 2, and 3 as "mild", grades 4, 5, and 6 as "moderate", and grades 7, 8, and 9 as "severe". Between these grades there is a small variation that is identified by the trained dermatologists, and which are taken into consideration to define the classification of the evaluated attribute (wrinkles/fine lines).
Clinical Efficacy Evaluations as Assessed by the Dermatologist on Day 56 | Day 56
  It is a clinical evaluation of the participant's face performed by a dermatologist according to a predefined scale. The attributes evaluated will be: wrinkles, and fine lines. A 10-point ordinal scale (0 to 9) developed by study site will be used where 0 = Absent and 9 = Numerous.Therefore, because it is an ordinal scale, the points in between do not have an established definition.
  Dermatologists have been trained to evaluate and classify grades 1, 2, and 3 as "mild", grades 4, 5, and 6 as "moderate", and grades 7, 8, and 9 as "severe". Between these grades there is a small variation that is identified by the trained dermatologists, and which are taken into consideration to define the classification of the evaluated attribute (wrinkles/fine lines).
Clinical Efficacy Evaluations as Assessed by the Dermatologist on Day 84 +/- 2 | Day 84 +/- 2
  It is a clinical evaluation of the participant's face performed by a dermatologist according to a predefined scale. The attributes evaluated will be: wrinkles, and fine lines. A 10-point ordinal scale (0 to 9) developed by study site will be used where 0 = Absent and 9 = Numerous.Therefore, because it is an ordinal scale, the points in between do not have an established definition.
  Dermatologists have been trained to evaluate and classify grades 1, 2, and 3 as "mild", grades 4, 5, and 6 as "moderate", and grades 7, 8, and 9 as "severe". Between these grades there is a small variation that is identified by the trained dermatologists, and which are taken into consideration to define the classification of the evaluated attribute (wrinkles/fine lines).

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielli Brianezi, Principal Investigator — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu